CLINICAL TRIAL: NCT02530047
Title: Phase 1 Study to Determine the Effects of Mesenchymal Stem Cells Secreting Interferon Beta in Patients With Advanced Ovarian Cancer
Brief Title: Mesenchymal Stem Cells (MSC) for Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0032; CA 136411 (Other: Ovarian Cancer SPORE Grant); NCI-2015-01504 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Epithelial ovarian cancer; Mesenchymal Stem Cells Secreting Interferon Beta; MSC-INFb; Questionnaires; Surveys
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Interferon-beta; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cells + Interferon Beta (MSC-INFβ) (Experimental): MSC-INFβ administered on an outpatient basis via intraperitoneal (IP) infusion. Starting dose: 10^5 MSC/kg once a week for 4 treatments. Up to 4 dose levels of MSC-INFβ tested. Symptom questionnaire completed once a week for 4 weeks.
  Interventions: Genetic: MSC-INFβ; Behavioral: Questionnaires

INTERVENTIONS:
Genetic: MSC-INFβ — MSC-INFβ administered on an outpatient basis via intraperitoneal (IP) infusion.
  Starting dose: 10^5 MSC/kg once a week for 4 treatments.
  Other Names: Mesenchymal stem cells with interferon beta
Behavioral: Questionnaires — Symptom questionnaire completed once a week for 4 weeks.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of human mesenchymal stem cells with interferon beta (MSC-INFb) that can be given to patients with ovarian cancer and to test the safety of the MSC-INFb.

This is an investigational study. MSC-INFb infusions for ovarian cancer is investigational.

Up to 21 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
MSCs are a type of stem cell that can be removed from bone marrow samples and grown into many different cell types that can be used to treat cancer. The MSCs used in this study were collected from healthy male donors and are stored in a laboratory at MD Anderson. The use of male cells will help us to detect the cells that are infused versus your own female cells.

The MSCs have been genetically changed in a laboratory at MD Anderson to add proteins called interferons. The MSCs will have genetic material introduced to them by a molecule called a plasmid that will help produce interferon beta. Interferons (IFNs) are proteins that may interfere with the growth of tumors. The MSCs will be grown in the laboratory and tested before they are given to you.

MSC-INFb Dose Levels:

If you are found eligible to take part in this study, you will be assigned to a dose level of MSC-INFb based on when you join this study. Up to 4 dose levels of MSC-INFb will be tested. Up to 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of MSC-INFb is found.

Your dose level may be lowered if you are not tolerating the MSC-INFb infusions. Your study doctor will discuss this with you.

MSC-INFb Administration:

About 1-2 weeks before your first MSC-INFb infusion, you will have an intraperitoneal (IP) catheter placed in your abdomen. A catheter is a sterile flexible tube that will be placed into your abdomen while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will receive a Patient Information Sheet that includes the definition of intraperitoneal therapy and information about the placement of the catheter and care of the catheter during the study. You will also be provided with a specific separate informed consent for the IP catheter placement by Interventional Radiology staff at MD Anderson.

One time a week for up to 4 weeks (up to 4 times total), you will receive the MSC-INFb infusions through the IP catheter. The length of time for the infusion will depend on the size of the tumor.

You will remain in the clinic for about 30 minutes for observation after each MSC-INFb infusion.

Study Tests:

About 1 week before your first MSC-INFb infusion:

* You will have a physical exam, including measurement of your weight and vital signs (blood pressure, heart rate, temperature, and breathing rate).
* Your medical history will be recorded.
* Blood (about 4 tablespoons each time) will be drawn for routine tests, to check your kidney and liver function, to check the status of the disease, and for INFb testing for comparison purposes. Blood tests may be repeated more frequently during the study if your doctor thinks it is needed.
* You will complete a symptom questionnaire. It should take about 10-15 minutes to complete.

About 1-2 weeks before your first MSC-INFb infusion, during the same procedure as the IP catheter placement, you will have a tumor biopsy to check the status of the disease. To collect a tumor biopsy, the affected area is numbed with anesthetic and a small amount of tissue is withdrawn with a large needle. A day or two before your tumor biopsy, blood (about 1 teaspoon) will be drawn to test clotting factors in your blood.

Once a week for 4 weeks, before each MSC-INFb infusion:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 4 tablespoons each time) will be drawn for routine tests, to check your kidney and liver function, to check the status of the disease and response to the infusion. °Blood tests may be repeated more frequently during the study if your doctor thinks it is needed.
* If you can become pregnant, you will have a blood or urine pregnancy test. If blood, it will be included in the routine blood draw listed above.
* Before the 1st, 2nd, and 3rd MSC-INFb infusion, you will complete a symptom questionnaire. It should take about 10-15 minutes each time to complete.
* Before each MSC-INFb infusion, up to 2 teaspoons of peritoneal fluid (if present) will be drawn through the catheter and stored in a laboratory at MD Anderson for future research related to this study.

Before your peritoneal fluid can be used for research, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee of doctors, researchers, and community members. The IRB is responsible for protecting study participants and making sure all research is safe and ethical.

Your samples will be given a code number. No identifying information will be directly linked to your samples. Only the researcher in charge of the bank will have access to the code numbers and be able to link the samples to you. This is to allow medical data related to the samples to be updated as needed.

About 22-26 days after your last MSC-INFb infusion:

* Blood (about 1 teaspoon) will be drawn to test clotting factors in your blood.
* You will have a tumor biopsy and the IP catheter will be removed. The tumor biopsy will be tested to determine if the MSC-INFb infusions had any effect on the tumor.
* You will have CT scans of the chest, abdomen, and pelvis to check the status of the disease. This may be repeated every 2 months for up to 12 months starting about 22-26 days after the last MSC-INFb infusion, if you doctor thinks it is needed.

Follow-Up Visits:

About 1 week after the last MSC-INFb infusion:

* You will have a physical exam, including measurement of your weight and vital signs.
* Blood (about 4 tablespoons) will be drawn about 1 week after the last MSC-INFb infusion for routine tests, to check your kidney and liver function, and to check the status of the disease and the response to the infusion. If your doctor thinks it is needed, blood (about 2 tablespoons each time) will be drawn at 44 days after the last MSC-INFb infusion and then once a month for 2 months to check the response to the infusions.
* You will complete a symptom questionnaire. It should take about 10-15 minutes to complete.

Length of Study:

You will be taken off study if the disease gets worse, if intolerable side effects occur, or your study doctor thinks it is in your best interest.

Long-Term Follow-Up:

For safety reasons, the U.S. Food and Drug Administration (FDA) requires that patients who receive infusions of stem cells treated with a gene transfer procedure must be followed have long-term follow-up for at least up to 15 years after receiving the gene transfer.

Once a year for Years 1-5 after the last MSC-INFb infusion:

* Blood (about 2-4 tablespoons each time) will be drawn for routine tests.
* You will have a physical exam, including measurement of your vital signs.
* You will complete a questionnaire that asks about your medical history (your general health, the status of any medical conditions, and any illnesses or hospitalizations that may have occurred). It should take about 15-30 minutes to complete.
* You will be asked if there have been any changes in your contact information.
* If necessary to check the status of the disease, you will have computed tomography (CT) scans and/or additional routine blood tests (about 1-2 tablespoons).

Once a year during Years 6-15 after the last MSC-INFb infusion, the research staff will contact you. Either over the phone, by email, or mail, you will fill out a questionnaire that asks about your medical history (your general health, the status of any medical conditions, and any illnesses or hospitalizations that may have occurred). The phone calls and questionnaires should take about 15-30 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 to 90 years in age with histologically documented diagnosis of epithelial ovarian cancer including serous papillary, endometrioid, mucinous, clear cell, poorly differentiated or mixed adenocarcinomas.
2. Patient must have recurrent epithelial ovarian cancer and may have received unlimited prior chemotherapeutic regimens for management of recurrent cancer.
3. Patients should have measurable disease as defined by RECIST 1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) that is accessible to biopsy.
4. Zubrod performance status of 0-1.
5. Absolute neutrophil count (ANC) > 1,000/mm3 and a platelet count > and a platelet count > 30,000/mm3.
6. Creatinine clearance > 50 mL/min (assessed by Cockcroft Gault estimation).
7. Bilirubin < 1.5 x upper limit of normal (unless Gilbert's syndrome), ALT or AST < 3 x upper limit of normal.
8. No evidence of significant cardiac or pulmonary dysfunction.
9. Patient must have a hemoglobin >/= 9 gm/dl (this may be achieved by transfusion if needed) obtained within 14 days before registration. If a patient receives packed red blood cell transfusion to achieve a hemoglobin level of >/= 9 gm/dl, the hemoglobin level needs to be stable (no drop by more than 1 gm/dl from the post-transfusion hemoglobin level) for at least 1 week.
10. Negative pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
11. Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months following last treatment.
12. Patient or patient's legal representative able to provide written informed consent.

Exclusion Criteria:

1. Patients receiving anti-cancer therapy within 21 days before MSC treatment.
2. Target lesion previously embolized, perfused, or irradiated without objective evidence of progression before start of therapy to be considered for response assessment.
3. Patients with uncontrolled symptomatic brain metastases. A scan to confirm absence of brain metastasis is not required.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic obstructive pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Symptomatic effusions due to pleural, pericardial, or peritoneal metastasis of epithelial ovarian cancer.
6. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, surgically treated Stage I or II cancer from which the patient is currently in complete remission (at least to 5 years), or any other cancer from which the patient has been disease-free for 5 years. Patients may have dual primaries of endometrial and ovarian cancer.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Mesenchymal Stem Cells-Interferon-β (MSC-IFNβ) | 5 weeks
  Maximum Tolerated Dose (MTD) is dose with posterior probability of dose limiting toxicities (DLTs) nearest to 30%, provided the lower bound of the 90% credible interval for the posterior probability of DLT does not exceed 30%. Dose limiting toxicities (DLTs) are those adverse events of grade 3 or 4 that occur up to 1 week after the last dose.
Correlation Between the Number of MSC-IFNβ Infused and the Production of Interferon-β and the Number of MSC-IFNβ Detected at the Tumor Sites Via Tumor Biopsy Pre- and Post-Treatment | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L. Olson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org